CLINICAL TRIAL: NCT03406507
Title: A Phase 3, Open-Label Study of ALXN1210 in Children and Adolescents With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Brief Title: A Study of Ravulizumab (ALXN1210) in Children and Adolescents With Paroxysmal Nocturnal Hemoglobinuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN1210-PNH-304; 2017-002820-26 (EudraCT Number)
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-02

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Ravulizumab; ALXN1210; Ultomiris; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ravulizumab (Experimental): Complement inhibitor treatment-naïve and eculizumab-experienced participants received ravulizumab.
  Interventions: Biological: Ravulizumab

INTERVENTIONS:
Biological: Ravulizumab — Single intravenous (IV) loading dose on Day 1, followed by regular IV maintenance dosing beginning on Day 15, based on weight.
  Other Names: ALXN1210; Ultomiris

SUMMARY:
The purpose of this study was to assess the pharmacokinetics (PK), pharmacodynamics (PD), safety, and efficacy of ravulizumab in pediatric participants with paroxysmal nocturnal hemoglobinuria (PNH).

DETAILED DESCRIPTION:
The study consists of a 4-week Screening Period, a 26-week Primary Evaluation Period, and an Extension Period of up to 4 years (with the exception of any country-specific mandates), whichever occurs first.

Efficacy and safety data are reported for the 26-week Primary Evaluation Period only. Analyses were conducted separately for complement inhibitor treatment-naïve participants and eculizumab-experienced participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants from birth up to <18 years of age and weighing ≥ 5 kilograms at the time of consent.
2. PNH diagnosis confirmed by documented high-sensitivity flow cytometry.
3. Presence of 1 or more of the following PNH-related signs or symptoms within 3 months of Screening: fatigue, hemoglobinuria, abdominal pain, shortness of breath (dyspnea), anemia, history of a major adverse vascular event (including thrombosis), dysphagia, or erectile dysfunction; or history of packed red blood cell transfusion due to PNH.
4. Lactate dehydrogenase (LDH) level ≥ 1.5 × upper limit of normal (ULN) for participants not being treated with eculizumab at screening and LDH level ≤ 1.5 × ULN for participants taking eculizumab.
5. Documented meningococcal vaccination not more than 3 years prior to dosing, and vaccination against Streptococcus pneumoniae and Haemophilus influenzae.
6. Female participants of childbearing potential must use highly effective contraception starting at screening and continuing until at least 8 months after the last dose of ravulizumab.

Exclusion Criteria:

1. History of bone marrow transplantation.
2. History of or ongoing major cardiac, pulmonary, renal, endocrine, or hepatic disease that, in the opinion of the investigator or sponsor, would preclude participation.
3. Unstable medical conditions (for example, myocardial ischemia, active gastrointestinal bleed, severe congestive heart failure, anticipated need for major surgery within 6 months of randomization, coexisting chronic anemia unrelated to PNH).
4. Females who are pregnant or breastfeeding or who have a positive pregnancy test at screening or Day 1.
5. Participation in another interventional clinical study or use of any experimental therapy within 30 days before initiation of study drug on Day 1 in this study or within 5 half-lives of that investigational product, whichever is greater.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (2):
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Milwaukee, Wisconsin
- Clinical Trial Site, Paris, France
- Clinical Trial Site, Utrecht, Netherlands
- Clinical Trial Site, Oslo, Norway
- Russia (2):
  - Clinical Trial Site, Moscow
  - Clinical Trial Site, Saint Petersburg
- United Kingdom (2):
  - Clinical Trial Site, Leeds
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Kulagin A, Chonat S, Maschan A, Bartels M, Buechner J, Punzalan R, Richards M, Ogawa M, Hicks E, Yu J, Baruchel A, Kulasekararaj AG. Pharmacokinetics, pharmacodynamics, efficacy, and safety of ravulizumab in children and adolescents with paroxysmal nocturnal hemoglobinuria: interim analysis of a phase 3, open-label study. Presented at the European Hematology Association 2021 Virtual Congress, June 9-17, 2021.
- [Derived] Chonat S, Kulagin A, Maschan A, Bartels M, Buechner J, Punzalan R, Richards M, Ogawa M, Hicks E, Yu J, Baruchel A, Kulasekararaj AG. Pharmacokinetics, pharmacodynamics, efficacy, and safety of ravulizumab in pediatric paroxysmal nocturnal hemoglobinuria. Blood Adv. 2024 Jun 11;8(11):2813-2824. doi: 10.1182/bloodadvances.2023012267. PMID 38551806

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen participants, from birth to < 18 years, were planned to be enrolled to ensure at least 10 evaluable participants would complete the 26-week Primary Evaluation Period. Participants were recruited from 9 sites across 6 countries (United States, United Kingdom, France, Netherlands, Russia, and Norway).
Groups:
- Treatment Naïve: Complement inhibitor treatment-naïve participants received weight-based doses of ravulizumab.
- Eculizumab Experienced: Eculizumab-experienced participants received weight-based doses of ravulizumab.
Period: Primary Evaluation Period
Arm/Group | Treatment Naïve | Eculizumab Experienced
Started | 5 | 8
Received at Least 1 Dose of Study Drug | 5 | 8
Completed | 5 | 8
Not Completed | 0 | 0
Period: Extension Period
Arm/Group | Treatment Naïve | Eculizumab Experienced
Started | 5 | 8
Received at Least 1 Dose of Study Drug | 5 | 8
Completed | 5 | 7
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis: all participants who received at least 1 dose of ravulizumab and had at least 1 efficacy assessment after the first infusion of ravulizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Naïve | Eculizumab Experienced | Total
Number analyzed (Participants) | 5 | 8 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at first infusion
  years | 14.4 (2.19) | 14.4 (3.07) | 14.4 (2.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 4 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Specific information pertaining to race and ethnicity undisclosed by Sponsor to ensure participant privacy.
  Participants
    Race - Undisclosed | 5 | 8 | 13
    Ethnicity - Undisclosed | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) Of Ravulizumab
Description: Blood samples for determination of ravulizumab Cmax were collected before and after administration of study drug at designated time points. Results are reported in micrograms/milliliter (μg/mL).
Time Frame: Week 1 (Day 1), Week 2 (Day 15), Week 10 (Day 71), and Week 18 (Day 127)
Population: Pharmacokinetic (PK): Participants enrolled into the study who received at least 1 dose of ravulizumab and who had evaluable interim PK data. The PK set was used for all PK analyses.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
μg/mL
  Day 1: End of Infusion | 725.40 (93.730) | 884.63 (170.842)
  Day 15: End of Infusion | 1161.60 (254.348) | 1612.50 (211.441)
  Day 71: End of Infusion: number analyzed (Participants) | 5 | 7
  Day 71: End of Infusion | 1402.00 (344.267) | 1581.43 (207.961)
  Day 127: End of Infusion | 1396.00 (403.770) | 1705.00 (164.751)

2. Primary Outcome: Trough Serum Concentration (Ctrough) Of Ravulizumab
Description: Blood samples for determination of ravulizumab Ctrough were collected before and after administration of study drug at designated time points. Trough serum concentration was measured at end of dosing interval at steady state. Results are reported in μg/mL.
Time Frame: Week 2 (Day 15), Week 10 (Day 71), Week 18 (Day 127), Week 26 (Day 183)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
μg/mL
  Day 15: Predose | 358.20 (51.978) | 452.25 (68.312)
  Day 71: Predose: number analyzed (Participants) | 5 | 7
  Day 71: Predose | 370.20 (134.267) | 521.00 (72.870)
  Day 127: Predose | 410.80 (215.503) | 554.88 (60.976)
  Day 183: Predose | 419.00 (191.921) | 565.63 (68.980)

3. Primary Outcome: Mean Accumulation Ratio For Cmax Of Ravulizumab Following The Last Maintenance Dose Relative To The First Maintenance Dose
Description: Blood samples for determination of ravulizumab accumulation ratio for Cmax were collected before and after administration of study drug at designated time points. The accumulation ratio was calculated as Cmax from the last maintenance dose (Week 18) divided by Cmax from the first maintenance dose (Week 2).
Time Frame: Week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
Ratio | 1.1995 (0.21038) | 1.0630 (0.06872)

4. Primary Outcome: Mean Accumulation Ratio For Ctrough Of Ravulizumab Following The Last Maintenance Dose Relative To The First Maintenance Dose
Description: Blood samples for determination of ravulizumab accumulation ratio for Ctrough were collected before and after administration of study drug at designated time points. The accumulation ratio was calculated as Ctrough from the last maintenance dose (Week 18) divided by Ctrough from the first maintenance dose (Week 2).
Time Frame: Week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 4 | 8
Ratio | 1.2208 (0.32490) | 1.0700 (0.09089)

5. Primary Outcome: Change In Free Complement Component C5 (C5) Concentrations Over Time
Description: Blood samples for determination of free C5 were collected before and after administration of study drug at designated time points.
Time Frame: Baseline, Weeks 2, 10, 18, and 26 (end of infusion)
Population: Pharmacodynamic: all participants who received at least 1 dose of ravulizumab and who had evaluable pharmacodynamic data.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
ug/mL
  Week 2 | -105.319 (17.1118) | 0.000 (0.0000)
  Week 10: number analyzed (Participants) | 5 | 6
  Week 10 | -105.310 (17.1139) | 0.003 (0.0052)
  Week 18 | -105.320 (17.1165) | 0.006 (0.0067)
  Week 26: number analyzed (Participants) | 5 | 7
  Week 26 | -105.320 (17.1184) | 0.006 (0.0070)

6. Primary Outcome: Change In Chicken Red Blood Cell (cRBC) Hemolytic Activity Over Time
Description: Blood samples for determination of cRBC hemolytic activity were collected before and after administration of study drug at designated time points.
Time Frame: Baseline, Weeks 2, 10, 18, and 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of hemolysis
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
percentage of hemolysis
  Week 2 | -93.12 (9.259) | 1.95 (2.816)
  Week 10: number analyzed (Participants) | 5 | 7
  Week 10 | -93.24 (9.241) | 3.97 (9.209)
  Week 18: number analyzed (Participants) | 4 | 8
  Week 18 | -96.93 (4.543) | 2.78 (5.673)
  Week 26: number analyzed (Participants) | 4 | 8
  Week 26 | -96.78 (4.816) | 7.03 (12.680)

7. Secondary Outcome: Percentage Change From Baseline At Week 26 In Lactate Dehydrogenase (LDH) Levels
Description: Blood and urine samples for determination of LDH levels were collected at designated time points. Baseline was defined as the average of all assessments analyzed by the central laboratory prior to first study drug administration.
Time Frame: Baseline, Week 26
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
Percent Change | -47.91 (52.716) | 4.65 (44.702)

8. Secondary Outcome: Percentage Of Participants Who Achieved Transfusion Avoidance (TA)
Description: Transfusion avoidance was defined as the proportion of participants who remained transfusion-free and did not require a transfusion according to protocol-specified guidelines. Point estimates and 2-sided 95% exact confidence intervals (CIs) were computed. Participants who withdrew from the study due to lack of efficacy during the Primary Evaluation Period were considered as non-responders and were counted in the group needing transfusion. For participants who withdrew from the study for any other reason during the Primary Evaluation Period, their data up to the time of withdrawal was used to assess TA.
Time Frame: Week 26
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
Percentage of Participants | 60.00 [14.66 to 94.73] | 100.00 [63.06 to 100.00]

9. Secondary Outcome: Change In Quality Of Life (QoL) From Baseline To Week 26
Description: Quality of life was measured by Pediatric Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Questionnaire (participants ≥ 5 years of age), a 13-item questionnaire that assesses fatigue and its impact upon daily activities and function over the preceding 7 days. Each item is scored on a 5-point scale, and total scores range from 0 to 52, with a higher score indicating better QoL. The scoring guideline for the Pediatric FACIT-Fatigue instrument was used to calculate a FACIT-Fatigue score. Changes from baseline in FACIT-Fatigue scores were summarized at baseline and at the study visits where this assessment was collected up to Day 183 (Week 26). At each study visit, the proportion of participants who showed an improvement of at least 3 points for the Pediatric FACIT-Fatigue scores were summarized by point estimates and 2-sided 95% exact CIs.
Time Frame: Baseline, Week 26
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
units on a scale | 3.40 (6.107) | 1.28 (5.235)

10. Secondary Outcome: Percentage Of Participants With Stabilized Hemoglobin At Week 26
Description: Stabilized hemoglobin was defined as avoidance of a ≥ 2 g/dL decrease in hemoglobin level from baseline in the absence of transfusion through Week 26. Point estimates and 2-sided 95% exact CIs were computed. Participants who withdrew from the study due to lack of efficacy during the Primary Evaluation Period were considered as non-responders and were counted in the group who did not meet the stabilized hemoglobin definition. For participants who withdrew from the study for any other reason during the Primary Evaluation Period, their data up to the time of withdrawal were used to assess stabilized hemoglobin.
Time Frame: Week 26
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
Percentage of Participants | 60.0 [14.66 to 94.73] | 75.0 [34.91 to 96.81]

11. Secondary Outcome: Percentage Change In Free Hemoglobin From Baseline To Week 26
Description: Percentage change from baseline in free hemoglobin was summarized at all study visits up to Day 183 (Week 26). Baseline was defined as the last non-missing assessment value prior to the first study drug infusion.
Time Frame: Baseline, Week 26
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
Percentage Change | 87.32 (226.816) | -15.29 (71.780)

12. Secondary Outcome: Percentage Of Participants With Breakthrough Hemolysis (BTH) At Week 26
Description: Breakthrough hemolysis was defined as at least one new or worsening symptom or sign of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, shortness of breath [dyspnea], anemia, major adverse vascular event [including thrombosis], dysphagia, or erectile dysfunction) in the presence of elevated LDH as follows: for participants who entered the study naïve to complement inhibitor treatment, elevated LDH ≥ 2 × the upper limit of normal (ULN) after prior LDH reduction to < 1.5 × ULN on therapy; for participants who entered the study stabilized on eculizumab treatment, elevated LDH ≥ 2 × ULN. Participants who withdrew from the study due to lack of efficacy during the Primary Evaluation Period were considered as non-responders and were counted in the group with BTH. For participants who withdrew from the study for any other reason during the Primary Evaluation Period, their data up to the time of withdrawal were used to assess BTH. No participants experienced BTH.
Time Frame: Week 26
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Naïve | Eculizumab Experienced
Number analyzed (Participants) | 5 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through End of Study (Up to Day 1610)
Arm/Group | Treatment Naïve | Eculizumab Experienced
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/8
Other Adverse Events (participants affected / at risk) | 4/5 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Naïve (N=5) | Eculizumab Experienced (N=8)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment Naïve (N=5) | Eculizumab Experienced (N=8)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 1 (4)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Electric shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Hyperbilirubinemia (Hepatobiliary disorders) | 1 (3) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
In growing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Administration site pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/1 (0) | 1/7 (1) — The N for this adverse event has been adjusted to the number of females in the study as it is a sex-specific event.
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Chromosomal deletion (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT03406507/Prot_002.pdf
  • Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT03406507/SAP_001.pdf